CLINICAL TRIAL: NCT03040076
Title: Testing if Reductions in Negative Affect Yield Decreased Emotional Eating Symptoms: A Cognitive Bias Intervention
Brief Title: Testing if Reductions in Negative Affect Yield Decreased Emotional Eating Symptoms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection suggested that more work was needed to validate the theoretical connections between the constructs of interest, before doing a treatment trial.
Sponsor: Florida State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016.19855
Record Dates: First submitted 2017-01-04; First posted 2017-02-02 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2016-12

CONDITIONS: Eating Disorder Symptom; Emotional Maladjustment; Negative Thoughts

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Treatment (Experimental): Intervention condition
  Interventions: Behavioral: Cognitive Bias Treatment
- Relaxation Condition (Active Comparator): Active control condition
  Interventions: Behavioral: Relaxation Condition

INTERVENTIONS:
Behavioral: Cognitive Bias Treatment — Two computerized tasks will be administered during four intervention sessions. During the first task, the Word Sentence Association Paradigm, participants see a threat or benign word and then an ambiguous sentence. Participants press one if they believe the word and sentence are related and two if they believe the word and sentence are not related. Participants are given feedback that they responded correctly if they state that a benign word is related to the sentence or they state that a threat word is not related to the sentence. The second task is the Ambiguous Scenarios Task. In each trial, an ambiguous scenario, ending in a benign word, appears on the screen. After the scenario is presented, participants respond to a comprehension question and are given feedback on their performance.
  Arms: Cognitive Bias Treatment
Behavioral: Relaxation Condition — Participants assigned to the active control group will complete four sessions of progressive muscle relaxation training. Two alternating relaxation scripts will be used. The scripts will be presented as Youtube videos with a blank black screen and will instruct participants to keep their eyes closed for the duration of the training. Participants will access the videos through Qualtrics to ensure that data can be gathered about their compliance. The relaxation scripts used in the present study will be modified versions of those currently being tested by other researchers utilizing cognitive bias modification paradigms. The relaxation training sessions will be matched to the length of the treatment condition and therefore will last approximately 30 minutes.
  Arms: Relaxation Condition

SUMMARY:
The purpose of this study to test a computerized treatment designed to help people with high levels of emotional eating, which is when people eat to cope with negative emotions and/or stressful situations. The investigators are interested in comparing two different ways of coping with negative emotions, relaxation training or training in how to think differently about such situations. Additionally, the researchers' study seeks to understand more about the psychological factors that may contribute to someone having difficulty with emotional eating.

DETAILED DESCRIPTION:
Emotional eating, or eating as a mechanism for coping with negative affect, is present across a spectrum of eating disorders and is associated with poor health outcomes, namely obesity. Research suggests that individuals with emotional eating experience urges to eat in response to multiple negative emotions, including anxiety, depression, and anger. While emotional eating is related to binge eating, it can be examined in a more dimensional fashion because it is not associated with a specific size criterion or a requirement of loss of control over eating. As such, emotional eating is a useful analog through which to understand mechanisms of binge eating and test the preliminary efficacy of treatment interventions. Interventions that target mechanisms of regulating negative affect may reduce both negative affect and emotional eating, increasing their transdiagnostic value. Research suggests that a large gap exists between the prevalence of psychopathology and access to psychological treatment, and this gap extends to individuals with eating disorders. A potential solution to these challenges is the use of computerized methodologies that may be easier to disseminate, allow for a gradient of treatment intensity, and do not rely upon training treatment providers. Computer-administered CBM interventions address the need for more easily disseminated treatments. CBM interventions are based in research suggesting that negative interpretation biases cause negative emotionality and subsequent symptom expression. Negative interpretation biases are the tendency to draw threatening conclusions about ambiguous information. Thus, CBM paradigms train people to make neutral or positive attributions about situations they would typically view through the lens of their negative biases. CBM interventions have been tested across a range of psychopathology, including anxiety disorders, depression, and anger, and using a variety of different bias modification techniques. Two recent CBM studies have been tested within the field of eating disorders. Although results were promising, both studies were marked by methodological limitations and neither addressed emotional eating specifically. The purpose of the present study is to test a CBM intervention designed to help individuals with elevated emotional eating improve their ability to regulate negative affect. In doing so, the investigators will determine if modifying the interpretation of ambiguous situations that would typically result in negative affect can reduce negative affect in individuals with high emotional eating. The researchers will in turn determine if those individuals have decreased food consumption under conditions that would otherwise elicit negative emotions. This project extends initial research on CBMs in eating disorders, as well as research suggesting that basic emotion regulation training can decrease emotional eating.

ELIGIBILITY:
Inclusion Criteria:

* Female between the ages of 18 and 45 years of age
* An emotional eating score more than one SD above the mean (>2.9) on the Dutch Eating Behavior Questionnaire (DEBQ) emotional eating scale (van Strien, Frijters, Bergers, & Defares, 1986).
* Regular computer and internet access
* Rate liking of vanilla frozen yogurt as a 6 or higher on a 10 point scale.

Exclusion Criteria:

* Body mass index (BMI; kg/m2) less than 18.5 (World Health Organization, 2000), given known cognitive impairments that can result from being underweight (Fowler et al., 2006).
* Current psychotic, manic, or substance use disorders, as these may interfere with their ability to cognitively engage in the intervention.
* Food allergies that would prevent consumption of vanilla frozen yogurt.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-05-03 (Actual)

PRIMARY OUTCOMES:
Change in Emotional Overeating Questionnaire Scores | Assessed at baseline (time zero), mid-treatment (8 days after baseline), and post-treatment (2 weeks after baseline).
  Emotional eating will be measured using the 6-item Emotional Overeating Questionnaire (EOQ; Masheb & Grilo, 2006), in which participants report on the frequency of eating in response to five negative emotions and one positive emotion. The instructions and item scaling will be modified to decrease the timeframe assessed from 28 days to 5 days, in order to be sensitive to changes during the present intervention. Each item will be assessed on a 5-point scale (0= no days to 5 = every day). Further, the instructions will be modified to not specifically reference eating an objectively large amount of food. This change is made in order to ensure consistency with how emotional eating is conceptualized in the literature (i.e., no specific size criterion). Change in scores at each of the time points will be used to determine symptom improvement.
Change in Positive and Negative Affect Schedule Scores | Assessed at baseline (time zero), mid-treatment (8 days after baseline), and post-treatment (2 weeks after baseline).
  Negative affect will be assessed using the negative affect scale of the Positive and Negative Affect Schedule (PANAS; Watson, Clark, & Tellegen, 1988), which is a 10-item measure of negative emotions on a scale of 1 ("very slightly or not at all) to 5 ("extremely"). The instructions can be modified as needed to reflect the desired timeframe of assessment (Watson et al., 1988) and therefore, we will instruct participants to consider the past five days.Change in scores at each of the time points will be used to determine symptom improvement.
Change in Word Sentence Association Paradigm Scores | Assessed at baseline (time zero), mid-treatment (8 days after baseline), and post-treatment (2 weeks after baseline).
  A modified version of the treatment condition Word Sentence Association Paradigm (WSAP; Amir & Taylor, 2012b; Beard & Amir, 2008; Hindash & Amir, 2012) will be used to assess interpretation bias. The ambiguous sentences will be distinct from those used in the bias modification program in order to allow for a more generalized assessment of change in biases. However, to permit an accurate assessment of changes in bias, the WSAP task will be the same at pre-, mid and post treatment. Scores on the WSAP task are calculated as the ratio of percent threatening to percent benign interpretations across the trials. Change in scores at each of the time points will be used to determine symptom improvement.

SECONDARY OUTCOMES:
Body Mass Index | Assessed at baseline (time zero).
  Body mass index (BMI) will be computed using participants' height, measured with a wall-mounted ruler, and weight, measured with an electronic scale.
Eating Pathology Symptoms Inventory | Assessed at baseline (time zero) and post-treatment (2 weeks after baseline).
  Eating disorder symptoms will be measured using the 8-item binge eating subscale of the Eating Pathology Symptoms Inventory (EPSI; Forbush et al., 2013), which measures features of binge eating (e.g., consumption of large quantities of food, mindless eating) on a 5-point Likert scale from "never" to "very often." The EPSI scale is designed to assess behavior over the past 28 days (Forbush et al., 2013); however, to be sensitive to the timeframe of the present study, the instructions will be modified to ask participants to consider the past week.
Depression and Anxiety Stress Scale | Assessed at baseline (time zero) and post-treatment (2 weeks after baseline).
  Depression, anxiety, and stress symptoms will be measured using the Depression and Anxiety Stress Scale (DASS; Lovibond & Lovibond, 1995a). The DASS is a 42-item measure that assesses such symptoms over the preceding week on a 0 to 3 scale from "did not apply to me at all" to "applied to me very much, or most of the time."
State-Trait Anger Expression Inventory, Second Edition | Assessed at baseline (time zero) and post-treatment (2 weeks after baseline).
  Anger symptoms will be measured using the trait anger scale of the State-Trait Anger Expression Inventory, Second Edition (STAXI-2; Spielberger, 1999). Only the trait scale will be used in the present study given our interest in assessing overall anger symptoms, not momentary anger levels, as a moderating variable. The trait scale consists of 10 items that assess frequency of anger a 4-point scale from "almost never" to "almost always," but is not measured across a specific timeframe (Spielberger & Reheiser, 2009).
Difficulties in Emotion Regulation Scale | Assessed at baseline (time zero) and post-treatment (2 weeks after baseline).
  Emotion dysregulation will be assessed using the Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004). The DERS is a 36-item measure of six aspects of emotion dysregulation; all items are measured on a 1 ("almost never") to 5 ("almost always") scale and are not anchored to a specific timeframe.
Visual Analogue Scale Ratings | Assessed at post-treatment (2 weeks after baseline).
  Before, during, and after a behavioral task designed to measure food consumption following stress, participants will complete Visual Analogue Scale (VAS; Rolls et al., 1992) ratings of hunger and fullness, as well as state affect (e.g., sad, anxious, frustrated, angry) by marking a 100-mm line (ends labeled from not at all to extremely).
Frozen Yogurt Consumption | Assessed at post-treatment (2 weeks after baseline).
  Food intake will be measured as the difference in weight of the frozen yogurt before and after the test meal (Geliebter et al., 2012) that is part of the behavioral stress task. The investigators will also record the time taken (out of fifteen minutes) participants used to consume the food.

OTHER OUTCOMES:
Psychological History | Assessed at baseline (time zero).
  Trained graduate students will administer modules of the Structured Clinical Interview for DSM 5 (SCID-5; First, Williams, Karg, & Spitzer, 2015), which will allow for an assessment of psychological treatment history and past/present eating disorder diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Keel, Ph.D., Principal Investigator — Department of Psychology, Florida State University
Locations (1):
- Eating Behaviors Research Clinic, Department of Psychology, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnow B, Kenardy J, Agras WS. The Emotional Eating Scale: the development of a measure to assess coping with negative affect by eating. Int J Eat Disord. 1995 Jul;18(1):79-90. doi: 10.1002/1098-108x(199507)18:13.0.co;2-v. PMID 7670446
- [Background] Van Strien T, Frijters JE, Bergers G, Defares PB. The Dutch Eating Behavior Questionnaire (DEBQ) for assessment of restrained, emotional, and external eating behavior. International Journal of Eating Disorders 5(2): 295-315, 1986.
- [Background] Masheb RM, Grilo CM. Emotional overeating and its associations with eating disorder psychopathology among overweight patients with binge eating disorder. Int J Eat Disord. 2006 Mar;39(2):141-6. doi: 10.1002/eat.20221. PMID 16231349
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Forbush KT, Wildes JE, Pollack LO, Dunbar D, Luo J, Patterson K, Petruzzi L, Pollpeter M, Miller H, Stone A, Bright A, Watson D. Development and validation of the Eating Pathology Symptoms Inventory (EPSI). Psychol Assess. 2013 Sep;25(3):859-78. doi: 10.1037/a0032639. Epub 2013 Jul 1. PMID 23815116
- [Background] Spielberger CD, Reheiser EC. Assessment of emotions: Anxiety, anger, depression, and curiosity. Applied Psychology: Health and Well-Being 1(3): 271-302, 2009.
- [Background] Amir N, Taylor CT. Interpretation training in individuals with generalized social anxiety disorder: a randomized controlled trial. J Consult Clin Psychol. 2012 Jun;80(3):497-511. doi: 10.1037/a0026928. Epub 2012 Jan 16. PMID 22250851
- [Background] Beard C, Amir N. A multi-session interpretation modification program: changes in interpretation and social anxiety symptoms. Behav Res Ther. 2008 Oct;46(10):1135-41. doi: 10.1016/j.brat.2008.05.012. Epub 2008 Jun 27. PMID 18675400
- [Background] Hindash AHC, Amir N. Negative interpretation bias in individuals with depressive symptoms. Cognitive Therapy and Research 36(5): 502-511, 2012.
- [Background] Amir N, Bomyea J, Beard C. The effect of single-session interpretation modification on attention bias in socially anxious individuals. J Anxiety Disord. 2010 Mar;24(2):178-82. doi: 10.1016/j.janxdis.2009.10.005. Epub 2009 Oct 27. PMID 19926442
- [Background] Cardi V, Esposito M, Bird G, Rhind C, Yiend J, Schifano S, Hirsch C, Treasure J. A preliminary investigation of a novel training to target cognitive biases towards negative social stimuli in Anorexia Nervosa. J Affect Disord. 2015 Dec 1;188:188-93. doi: 10.1016/j.jad.2015.08.019. Epub 2015 Aug 28. PMID 26363616
- [Background] Hayes S, Hirsch CR, Krebs G, Mathews A. The effects of modifying interpretation bias on worry in generalized anxiety disorder. Behav Res Ther. 2010 Mar;48(3):171-8. doi: 10.1016/j.brat.2009.10.006. Epub 2009 Oct 14. PMID 19857859
- [Background] Hirsch CR, Hayes S, Mathews A. Looking on the bright side: accessing benign meanings reduces worry. J Abnorm Psychol. 2009 Feb;118(1):44-54. doi: 10.1037/a0013473. PMID 19222313
- [Background] Rolls BJ, Andersen AE, Moran TH, McNelis AL, Baier HC, Fedoroff IC. Food intake, hunger, and satiety after preloads in women with eating disorders. Am J Clin Nutr. 1992 Jun;55(6):1093-103. doi: 10.1093/ajcn/55.6.1093. PMID 1595580
- [Background] Kirschbaum C, Pirke KM, Hellhammer DH. The 'Trier Social Stress Test'--a tool for investigating psychobiological stress responses in a laboratory setting. Neuropsychobiology. 1993;28(1-2):76-81. doi: 10.1159/000119004. PMID 8255414
- [Background] Geliebter A, Gibson CD, Hernandez DB, Atalayer D, Kwon A, Lee MI, Mehta N, Phair D, Gluck ME. Plasma cortisol levels in response to a cold pressor test did not predict appetite or ad libitum test meal intake in obese women. Appetite. 2012 Dec;59(3):956-9. doi: 10.1016/j.appet.2012.08.025. Epub 2012 Sep 13. PMID 22983369
- [Background] Fowler L, Blackwell A, Jaffa A, Palmer R, Robbins TW, Sahakian BJ, Dowson JH. Profile of neurocognitive impairments associated with female in-patients with anorexia nervosa. Psychol Med. 2006 Apr;36(4):517-27. doi: 10.1017/S0033291705006379. Epub 2005 Dec 1. PMID 16318655
- [Background] Kirschbaum, C. (2010). Trier social stress test. In I.P. Stolerman (Ed.), Encyclopedia of Psychopharmacology (pp. 1346-1346). Germany: Springer Berlin Heidelberg.
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] First, M.B., Williams, J.B.W., Karg, R.S., & Spitzer, R.L (2015). Structured clinical interview for DSM-5 disorders. Arlington, VA: American Psychiatric Publishing.
- [Background] Lovibond, S. H., & Lovibond, P. F. (1995). Manual for the Depression Anxiety Stress Scales (DASS). Sydney, Australia: Psychology Foundation of Australia.
- [Background] Spielberger, C. D. (1999). State-Trait Anger Expression Inventory-2: Professional Manual. Lutz, FL: Psychological Assessment Resources.
- [Background] Habhab S, Sheldon JP, Loeb RC. The relationship between stress, dietary restraint, and food preferences in women. Appetite. 2009 Apr;52(2):437-44. doi: 10.1016/j.appet.2008.12.006. Epub 2008 Dec 24. PMID 19135112
- [Background] Laitinen J, Ek E, Sovio U. Stress-related eating and drinking behavior and body mass index and predictors of this behavior. Prev Med. 2002 Jan;34(1):29-39. doi: 10.1006/pmed.2001.0948. PMID 11749094
- [Background] Duarte C, Pinto-Gouveia J. Returning to emotional eating: the emotional eating scale psychometric properties and associations with body image flexibility and binge eating. Eat Weight Disord. 2015 Dec;20(4):497-504. doi: 10.1007/s40519-015-0186-z. Epub 2015 Feb 27. PMID 25721943
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Hart LM, Granillo MT, Jorm AF, Paxton SJ. Unmet need for treatment in the eating disorders: a systematic review of eating disorder specific treatment seeking among community cases. Clin Psychol Rev. 2011 Jul;31(5):727-35. doi: 10.1016/j.cpr.2011.03.004. Epub 2011 Mar 23. PMID 21501580
- [Background] Hallion LS, Ruscio AM. A meta-analysis of the effect of cognitive bias modification on anxiety and depression. Psychol Bull. 2011 Nov;137(6):940-58. doi: 10.1037/a0024355. PMID 21728399
- [Background] Amir N, Taylor CT. Combining computerized home-based treatments for generalized anxiety disorder: an attention modification program and cognitive behavioral therapy. Behav Ther. 2012 Sep;43(3):546-59. doi: 10.1016/j.beth.2010.12.008. Epub 2011 May 30. PMID 22697443
- [Background] Hawkins KA, Cougle JR. Effects of interpretation training on hostile attribution bias and reactivity to interpersonal insult. Behav Ther. 2013 Sep;44(3):479-88. doi: 10.1016/j.beth.2013.04.005. Epub 2013 Apr 19. PMID 23768674
- [Background] Mathews A, Ridgeway V, Cook E, Yiend J. Inducing a benign interpretational bias reduces trait anxiety. J Behav Ther Exp Psychiatry. 2007 Jun;38(2):225-36. doi: 10.1016/j.jbtep.2006.10.011. Epub 2006 Dec 1. PMID 17141179
- [Background] Salemink E, van den Hout M, Kindt M. Effects of positive interpretive bias modification in highly anxious individuals. J Anxiety Disord. 2009 Jun;23(5):676-83. doi: 10.1016/j.janxdis.2009.02.006. Epub 2009 Feb 14. PMID 19272750
- [Background] Yiend J, Parnes C, Shepherd K, Roche MK, Cooper M. Negative self-beliefs in eating disorders a cognitive-bias-modification study. Clinical Psychological Science, 2(6): 756-766, 2014.
- [Background] Svaldi J, Tuschen-Caffier B, Trentowska M, Caffier D, Naumann E. Differential caloric intake in overweight females with and without binge eating: effects of a laboratory-based emotion-regulation training. Behav Res Ther. 2014 May;56:39-46. doi: 10.1016/j.brat.2014.02.008. Epub 2014 Mar 7. PMID 24650627
- [Background] Gratz KL, Roemer L. Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment 26(1): 41-54, 2004.